CLINICAL TRIAL: NCT01894113
Title: Prospective, Randomised Multicenter Study Comparing Transbronchial Forceps Biopsy With Cryobiopsy in Interstitial Lung Disease
Brief Title: Prospective, Randomised Multicenter Study Comparing the Efficacy of Transbronchial Forceps Biopsy With Cryobiopsy to Diagnose Interstitial Lung Disease.
Acronym: TRABIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Boeckeler, Michael, Dr. med. Michael Böckeler, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: TBB2010
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Interstitial Lung Disease
Keywords: interstitial lung disease; transbronchial biopsy; cryobiopsy
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- transbronchial forceps lung biopsy (Active Comparator): transbronchial lung biopsy forceps
  Interventions: Procedure: transbronchial lung biopsy
- transbronchail cryo lung biopsy (Active Comparator): transbronchial lungbiopsy with cryoprobe
  Interventions: Procedure: transbronchial lung biopsy

INTERVENTIONS:
Procedure: transbronchial lung biopsy

SUMMARY:
The use of cryoprobes improves the diagnostic yield in transbronchial biopsies compared to forceps biopsies to diagnose an interstitial lung disease

DETAILED DESCRIPTION:
Endoscopic biopsy currently plays only a minor role for the diagnosis of interstitial lung disease. However, in some cases obtaining lung tissue is necessary to establish a final diagnosis. The current standard procedure is transbronchial forceps biopsy - if not sufficient: surgical lung biopsy. Transbronchial lung biopsy bears essential limitations however:

* Small tissue sample
* Limited evaluability of the material caused by forceps-induced crush artifacts

In cryobiopsy the cryoprobe´s tip is being cooled and thereby cools the surrounding tissue to approximately minus 89 degrees Celsius. Subsequently, the frozen probe is retracted with the frozen tissue being attached onto the frozen probe's tip. When applied in the central airways, cryobiopsy proved to deliver large specimens of good quality, which may exceed forceps biopsies in terms of diagnostic yield. Pilot studies on transbronchial cryobiopsy showed that same advantages as seen in the endobronchial use.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical indications for biopsy of interstitial lung disease
2. Age over 18 years
3. Signed consent

Exclusion Criteria:

1. Risk of bleeding / ongoing anticoagulation
2. Oxygen saturation <90% - despite delivery of 2l oxygen / min
3. Underlying cardiac disease (unstable angina, myocardial infarction during the last month, congestive heart failure)
4. Pulmonary hypertension, PAP sys> 50mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Diagnostic value of each biopsy procedure. It will be identified, how often biopsy contributed to the final diagnosis. | 24 months

SECONDARY OUTCOMES:
Differences in the final diagnosis | 24 Months

OTHER OUTCOMES:
Bleeding None, Mild degree (suction <= 3min), Moderate (extraction> 3min), Severe (intervention: tamponade, surgery) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Hetzel, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

REFERENCES:
- [Derived] Hetzel J, Eberhardt R, Petermann C, Gesierich W, Darwiche K, Hagmeyer L, Muche R, Kreuter M, Lewis R, Ehab A, Boeckeler M, Haentschel M. Bleeding risk of transbronchial cryobiopsy compared to transbronchial forceps biopsy in interstitial lung disease - a prospective, randomized, multicentre cross-over trial. Respir Res. 2019 Jul 5;20(1):140. doi: 10.1186/s12931-019-1091-1. PMID 31277659